CLINICAL TRIAL: NCT02499146
Title: A PHASE 1 OPEN-LABEL PHARMACOKINETICS STUDY OF PALBOCICLIB, A CYCLIN-DEPENDENT KINASE 4 AND 6 (CDK4/6) INHIBITOR, IN POSTMENOPAUSAL CHINESE WOMEN WITH ER (+), HER2 (-) ADVANCED BREAST CANCER
Brief Title: Palbociclib Pharmacokinetics Study In Postmenopausal Chinese Women With ER (+), HER2 (-) Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A5481019; NCT02499146 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Advanced Breast Cancer
Keywords: Palbociclib; PD-0332991; pharmacokinetics; breast cancer patients; Chinese
MeSH Terms: interventions — palbociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 1 (Experimental): Combination therapy of palbociclib and letrozole
  Interventions: Drug: Palbociclib; Drug: Letrozole

INTERVENTIONS:
Drug: Palbociclib — 125 mg orally once daily with food on Day 1 to Day 21 followed by 7 days off treatment in a 28-day cycle
Drug: Letrozole — 2.5 mg , orally once daily (continuously)

SUMMARY:
As part of the global clinical development program for Palbociclib, studies are planned in cancer patients in China. An assessment of Palbociclib pharmacokinetics in Chinese patients, as required by the Chinese Health Authorities, is therefore warranted. In addition, safety and efficacy will be also evaluated.

The single and multiple 125 mg oral dose pharmacokinetics of Palbociclib will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* ER(+), HER2(-), postmenopausal adult (ages 18-65 years, inclusive) Chinese women with proven diagnosis of adenocarcinoma of the breast with evidence locoregionally recurrent or metastatic disease not amenable to resection or radiation therapy with curative intent and for whom chemotherapy is not clinically indicated.

  a. Postmenopausal women: i. Prior bilateral surgical oophorectomy; or ii. Medically confirmed post-menopausal status defined as spontaneous cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause b. Documentation of histologically or cytologically confirmed diagnosis of: i. ER(+) breast cancer. c. Documentation of HER2(-) breast cancer. d. Previously untreated with any systemic anti cancer therapy for their locoregionally recurrent or metastatic ER+ disease.
* Measurable disease as defined per RECIST v.1.1 or bone-only disease. - Tumor lesions previously irradiated or subjected to other locoregional therapy will only be deemed measurable if disease progression at the treated site after completion of therapy is clearly documented.

Exclusion Criteria:

* HER2-positive tumor as defined by documentation of erbB-2 gene amplification by FISH (as defined by a HER2/CEP17 ratio ≥2) or chromogenic in situ hybridization (CISH, as defined by the manufacturer's kit instruction) or documentation of HER2 overexpression by IHC (defined as IHC3+, or IHC2+ with FISH or CISH confirmation) based on local laboratory results
* Patients with advanced, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term (including patients with massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver involvement).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2024-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- China (7):
  - Beijing Cancer Hospital/Oncology department, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong General Hospital/Department of Breast Surgery, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The first hospital of jilin university, Changchun, Jilin
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Yu Y, Sun W, Liu Y, Wang D. Pharmacodynamic Modeling of CDK4/6 Inhibition-Related Biomarkers and the Characterization of the Relationship Between Biomarker Response and Progression-Free Survival in Patients With Advanced Breast Cancer. J Clin Pharmacol. 2022 Mar;62(3):376-384. doi: 10.1002/jcph.1971. Epub 2021 Nov 16. PMID 34554584
- [Derived] Xu B, Li H, Zhang Q, Sun W, Yu Y, Li W, Wang S, Liao N, Shen P, Liu Y, Huang Y, Linn C, Zhao H, Jiang J, Wang D. Pharmacokinetics, safety, activity, and biomarker analysis of palbociclib plus letrozole as first-line treatment for ER+/HER2- advanced breast cancer in Chinese women. Cancer Chemother Pharmacol. 2021 Jul;88(1):131-141. doi: 10.1007/s00280-021-04263-9. Epub 2021 Apr 9. PMID 33835229
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481019&StudyName=Palbociclib%20%28PD-0332991%29%20Pharmacokintetics%20Study%20In%20Postmenopausal%20Chinese%20Women%20With%20ER%20%28+%29%2C%20HER2%20%28-%29%20Advanced%20Breast%20Cancer%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Palbociclib + Letrozole: Participants received a single dose of palbociclib 125 milligrams (mg) orally on Day 1 during the 5-day lead-in phase and received once daily (QD) from Day 1 to Day 21 (followed by 7 days off-treatment) during each 28-day treatment cycle. A treatment cycle was defined as 28 days in duration and Cycle 1 started on Day 6 of lead-in phase as Cycle 1 Day 1. Letrozole 2.5 mg was administered orally QD from Days 1 to 5 during the 5-day lead-in phase and from Days 1 to 28 during each 28-day treatment cycle.
Period: Overall Study
Arm/Group | Palbociclib + Letrozole
Started | 26
Completed | 0
Not Completed | 26
Not completed — Global deterioration of health status | 1
Not completed — Objective progression or relapse | 20
Not completed — Other | 2
Not completed — Participant refused continued treatment for reason other than adverse event | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study medication.
Groups:
- Palbociclib + Letrozole: Participants received palbociclib 125 milligrams (mg) orally once daily (QD) on Day 1 during the 5-day lead-in phase and from Day 1 to Day 21 (followed by 7 days off-treatment) during each treatment cycle. A treatment cycle was defined as 28 days in duration and Cycle 1 was started with Day 6 of lead-in phase as Cycle 1 Day 1. Letrozole 2.5 mg was administered orally QD from Days 1 to 5 during the 5-day lead-in phase and from Days 1 to 28 during each 28-day treatment cycle.
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 26

OUTCOME MEASURES:

1. Primary Outcome: Single-dose Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) for Palbociclib
Description: Cmax of palbociclib in the single-dose part (lead-in phase) was observed directly from data.
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, 24, 48, 72, 96 and 120 hours post dose
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Palbociclib + Letrozole: Participants received a single dose of palbociclib 125 mg orally on Day 1 during the 5-day lead-in phase and received once QD from Day 1 to Day 21 (followed by 7 days off-treatment) during each 28-day treatment cycle. A treatment cycle was defined as 28 days in duration and Cycle 1 started on Day 6 of lead-in phase as Cycle 1 Day 1. Letrozole 2.5 mg was administered orally QD from Days 1 to 5 during the 5-day lead-in phase and from Days 1 to 28 during each 28-day treatment cycle.
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
nanograms per milliliter (ng/mL) | 82.14 (25)

2. Primary Outcome: Single-dose PK: Time to Reach Maximum Plasma Concentration (Tmax) for Palbociclib
Description: Tmax for palbociclib in the single-dose part (lead-in phase) was observed directly from data as time of first occurrence.
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, 24, 48, 72, 96 and 120 hours post dose
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose part.
Measure: Median (Full Range); unit: hours
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
hours | 7.94 [3.97 to 10.0]

3. Primary Outcome: Single-dose PK: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time 0 to the Time 10 Hours (AUC10) for Palbociclib
Description: AUC10 for palbociclib in the single-dose part (lead-in phase) was obtained by linear/log trapezoidal method.
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, and 10 hours post dose
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
nanograms*hour per milliliter (ng*hr/mL) | 498.3 (28)

4. Primary Outcome: Single-dose PK: AUC From Time 0 to the Time 24 Hours (AUC24) for Palbociclib
Description: AUC24 is AUCtau, where the dosing interval (tau) is 24 hours. AUC24 in the single-dose part (lead-in phase) for palbociclib was obtained by linear/log trapezoidal method.
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, and 24 hours post dose
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
ng*hr/mL | 1217 (22)

5. Primary Outcome: Single-dose PK: AUC From Time 0 to the Time of Last Quantifiable Concentration (AUClast) for Palbociclib
Description: AUClast for palbociclib in the single-dose part (lead-in phase) was obtained by linear/log trapezoidal method.
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, 24, 48, 72, 96 and 120 hours post dose
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
ng*hr/mL | 2308 (27)

6. Primary Outcome: Single-dose PK: AUC From Time 0 Extrapolated to Infinite Time (AUCinf) for Palbociclib
Description: AUCinf for palbociclib in the single-dose part (lead-in phase) was calculated as AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis and kel was the rate constant for terminal phase obtained by linear regression of the log-linear concentration-time curve.
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, 24, 48, 72, 96 and 120 hours post dose
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
ng*hr/mL | 2386 (27)

7. Primary Outcome: Single-dose PK: Rate Constant for Terminal Phase (Kel) for Palbociclib
Description: Kel for palbociclib in the single-dose part (lead-in phase) was obtained by linear regression of the log-linear concentration-time curve.
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, 24, 48, 72, 96 and 120 hours post dose
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose part.
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
per hour | 0.03006 (0.00420)

8. Primary Outcome: Single-dose PK: Mean Residence Time (MRT) for Palbociclib
Description: MRT for palbociclib in the single-dose part (lead-in phase) was calculated as AUMCinf/AUCinf, where AUMCinf was area under the first moment curve from time 0 to infinity.
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, 24, 48, 72, 96 and 120 hours post dose
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose part.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
hours | 34.42 (4.32)

9. Primary Outcome: Single-dose PK: Terminal Half-Life (t1/2) for Palbociclib
Description: t1/2 for palbociclib in the single-dose part (lead-in phase) was calculated as Loge(2)/kel.
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, 24, 48, 72, 96 and 120 hours post dose
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose part.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
hours | 23.46 (3.14)

10. Primary Outcome: Single-dose PK: Apparent Oral Clearance (CL/F) for Palbociclib
Description: CL/F for palbociclib in the single-dose part (lead-in phase) was calculated as Dose/AUCinf.
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, 24, 48, 72, 96 and 120 hours post dose
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/hr)
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
liters per hour (L/hr) | 52.40 (27)

11. Primary Outcome: Single-dose PK: Apparent Volume of Distribution (Vz/F) for Palbociclib
Description: Vz/F for palbociclib in the single-dose part (lead-in phase) was calculated as Dose/(AUCinf * kel).
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, 24, 48, 72, 96 and 120 hours post dose
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
liters | 1758 (21)

12. Primary Outcome: Multiple-dose PK: Maximum Plasma Concentration at Steady State (Css,Max) for Palbociclib
Description: Css,max of palbociclib in the multiple-dose part (Cycle 1) was observed directly from data.
Time Frame: Cycle 1: pre-dose on Day 19, Day 20, Day 21, and 2, 4, 6, 8, 10, 24, 48, 72, 96, 120 hours post dose on Day 21
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the multiple-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 24
ng/mL | 139.7 (28)

13. Primary Outcome: Multiple-dose PK: Minimum Plasma Concentration at Steady State (Css,Min) for Palbociclib
Description: Css,min of palbociclib in the multiple-dose part (Cycle 1) was observed directly from data.
Time Frame: Cycle 1: pre-dose on Day 19, Day 20, Day 21, and 2, 4, 6, 8, 10, 24, 48, 72, 96, 120 hours post dose on Day 21
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the multiple-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 24
ng/mL | 67.55 (46)

14. Primary Outcome: Multiple-dose PK: AUC Within a Dosing Interval of Tau (=24 Hours) at Steady State (AUCss,Tau) for Palbociclib
Description: AUCss,tau of palbociclib in the multiple-dose part (Cycle 1) was determined by linear/log trapezoidal method.
Time Frame: Cycle 1: pre-dose on Day 19, Day 20, Day 21, and 2, 4, 6, 8, 10, and 24 hours post dose on Day 21
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the multiple-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 24
ng*hr/mL | 2501 (29)

15. Primary Outcome: Multiple-dose PK: Average Plasma Concentration at Steady State (Css,av) for Palbociclib
Description: Css,av of palbociclib in the multiple-dose part (Cycle 1) was calculated as AUCss,tau/tau, where tau was 24 hours.
Time Frame: Cycle 1: pre-dose on Day 19, Day 20, Day 21, and 2, 4, 6, 8, 10, and 24 hours post dose on Day 21
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the multiple-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 24
ng/mL | 104.2 (29)

16. Primary Outcome: Multiple-dose PK: Time to Reach Maximum Plasma Concentration at Steady State (Tss,Max) for Palbociclib
Description: Tss,max of palbociclib in the multiple-dose part (Cycle 1) was observed directly from data as time of first occurrence within tau (=24 hours) at steady state.
Time Frame: Cycle 1: pre-dose on Day 19, Day 20, Day 21, and 2, 4, 6, 8, 10, and 24 hours post dose on Day 21
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the multiple-dose part.
Measure: Median (Full Range); unit: hours
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 24
hours | 6.05 [3.97 to 10.0]

17. Primary Outcome: Multiple-dose PK: Vz/F for Palbociclib
Description: Vz/F of palbociclib in the multiple-dose part (Cycle 1) was calculated as Dose/(AUCss,tau * kel), where AUCss,tau was the AUC within a dosing interval of tau (=24 hours) at steady state and kel was the terminal phase rate constant following multiple-dose calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Cycle 1: pre-dose on Day 19, Day 20, Day 21, and 2, 4, 6, 8, 10, 24, 48, 72, 96, 120 hours post dose on Day 21
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest and a well characterized terminal phase in the multiple-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 23
Liters | 1910 (29)

18. Primary Outcome: Multiple-dose PK: t1/2 for Palbociclib
Description: t1/2 of palbociclib in the multiple-dose part (Cycle 1) was calculated as ln (2)/kel, where kel was the terminal phase rate constant following multiple-dose calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Cycle 1: pre-dose on Day 19, Day 20, Day 21, and 2, 4, 6, 8, 10, 24, 48, 72, 96, 120 hours post dose on Day 21
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest and a well characterized terminal phase in the multiple-dose part .
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 23
hours | 27.26 (3.19)

19. Primary Outcome: Multiple-dose PK: CL/F for Palbociclib
Description: CL/F of palbociclib in the multiple-dose part (Cycle 1) was calculated as Dose/AUCss,tau, where AUCss,tau was the AUC within a dosing interval of tau (=24 hours) at steady state.
Time Frame: Cycle 1: pre-dose on Day 19, Day 20, Day 21, and 2, 4, 6, 8, 10, and 24 hours post dose on Day 21
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the multiple-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 24
L/hr | 49.97 (29)

20. Primary Outcome: Multiple-dose PK: Peak to Trough Fluctuation at Steady State (PTF) for Palbociclib
Description: PTF of palbociclib in the multiple-dose part (Cycle 1) was determined as (Css,max - Css,min)/Css,av. Css,max and Css,min were observed directly from data while Css,av was calculated as AUCss,tau/tau, where tau was 24 hours.
Time Frame: Cycle 1: pre-dose on Day 19, Day 20, Day 21, and 2, 4, 6, 8, 10, 24, 48, 72, 96, 120 hours post dose on Day 21
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the multiple-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 24
ratio | 0.6652 (27)

21. Primary Outcome: Observed Accumulation Ratio (Rac) for Palbociclib
Description: Rac of palbociclib was determined as AUCss,tau/AUCsd,tau, where AUCss,tau (tau=24 hours) was from multiple-dose part (Cycle 1) and AUCsd,tau was AUC24 from single-dose part (lead-in phase).
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, and 24 hours post dose; Cycle 1: pre-dose on Day 19, Day 20, Day 21, and 2, 4, 6, 8, 10, and 24 hours post dose on Day 21
Population: All enrolled and treated participants who had at least 1 PK parameter of primary interest in the single-dose and multiple-dose part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 24
ratio | 2.042 (27)

22. Primary Outcome: Steady State Accumulation Ratio (Rss) for Palbociclib
Description: Rss of palbociclib was calculated as AUCss,tau/AUCinf, where AUCss,tau (tau=24 hours) was from multiple-dose part (Cycle 1) and AUCinf was from single-dose part (lead-in phase).
Time Frame: Lead-in phase: Day 1 pre-dose, 2, 4, 6, 8, 10, 24, 48, 72, 96 and 120 hours post dose; Cycle 1: pre-dose on Day 19, Day 20, Day 21, and 2, 4, 6, 8, 10, 24 hours post dose on Day 21
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 24
ratio | 1.036 (26)

23. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or increasing in severity on or after the first dose of investigational product administration. AEs included both SAEs and non-serious AEs. Causality to study treatment was determined by the investigator.
Time Frame: From first dose of study medication up to 28 days after last dose of study medication (up to maximum of 475 weeks, maximum treatment exposure = 471 weeks)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
Participants
  Treatment-emergent AEs (all causalities) | 26
  Treatment-emergent AEs (treatment-related) | 26
  Treatment-emergent SAEs (all causalities) | 4
  Treatment-emergent SAEs (treatment-related) | 1

24. Secondary Outcome: Number of Participants With Treatment-Emergent AEs by Maximum National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or increasing in severity on or after the first dose of investigational product administration. AEs included both SAEs and non-serious AEs. Causality to study treatment was determined by the investigator. AEs were graded by NCI CTCAE version 4.0: Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: as for outcome 23
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
Participants
  Grade 1 | 0
  Grade 2 | 5
  Grade 3 | 16
  Grade 4 | 5
  Grade 5 | 0

25. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: The number of participants with the following laboratory test abnormalities meeting any of the Grades 1 to 4 criteria per the NCI CTCAE (version 4.0) is summarized: anemia, lymphopenia, neutropenia, platelet count decreased, white blood cell (WBC) decreased, alanine aminotransferase (ALT) increased, alkaline phosphatase increased, aspartate aminotransferase (AST) increased, bilirubin (total) increased, creatinine increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, and hyponatremia. Grade 1=mild, Grade 2=moderate, Grade 3=severe and Grade 4=life-threatening. One participant might had more than 1 laboratory test abnormality.
Time Frame: as for outcome 23
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
Participants
  Anemia | 23
  Lymphopenia | 19
  Neutropenia | 26
  Platelet count decreased | 20
  WBC decreased | 25
  ALT increased | 11
  Alkaline phosphatase increased | 12
  AST increased | 18
  Bilirubin (total) increased | 4
  Creatinine increased | 25
  Hypercalcemia | 1
  Hyperglycemia | 10
  Hyperkalemia | 0
  Hypermagnesemia | 2
  Hypernatremia | 6
  Hypoalbuminemia | 11
  Hypocalcemia | 11
  Hypoglycemia | 0
  Hypokalemia | 6
  Hypomagnesemia | 5
  Hyponatremia | 6

26. Secondary Outcome: Number of Participants Meeting the Categorical Summarization Criteria for QTcF and QTcB Parameters
Description: QT interval (time from electrocardiogram [ECG] Q wave and the end of the T wave corresponding to electrical systole) corrected for heart rate using Fridericia's formula was QTcF and QT interval corrected for heart rate using Bazett's formula was QTcB. Categorical summarization criteria for QTcF and QTcB were as follows: 1) maximum absolute value of <450 milliseconds (msec), >=450 to <=480 msec, >=481 to <=500 msec, or >=500 msec; 2) maximum increase from baseline of <30 msec, >=30 to <60 msec, or >=60 msec. One participant could be reported under more than 1 categorical summarization criteria for QTcF and QTcB Parameters.
Time Frame: as for outcome 23
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
Participants
  Maximum QTcF <450 msec | 21
  Maximum QTcF >=450 to <=480 msec | 4
  Maximum QTcF >=481 to <=500 msec | 1
  Maximum QTcF >500 msec | 0
  Maximum increase in QTcF <30 msec | 17
  Maximum increase in QTcF >=30 to <60 msec | 9
  Maximum increase in QTcF >=60 msec | 0
  Maximum QTcB <450 msec | 9
  Maximum QTcB >=450 to <=480 msec | 16
  Maximum QTcB >=481 to <=500 msec | 0
  Maximum QTcB >500 msec | 1
  Maximum increase in QTcB <30 msec | 16
  Maximum increase in QTcB >=30 to <60 msec | 9
  Maximum increase in QTcB >=60 msec | 1

27. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from Cycle 1 Day 1 (C1D1) to date of first documentation of disease progression (PD) or death due to any cause, whichever occurred first. Documentation of progression was by objective disease assessment as defined by the Response Evaluation Criteria in Solid Tumor (RECIST) (version 1.1). PD was defined as a >=20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 millimeter (mm); or unequivocal progression of pre-existing lesions for non-target disease; or appearance of new unequivocal malignant lesions. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: From C1D1 to date of first documentation of PD or death due to any cause, whichever occurred first (up to maximum of 471 weeks of treatment exposure)
Population: Efficacy analysis set included all enrolled participants who started the treatment of Cycle 1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
Months | 18.6 [6.5 to 27.7]

28. Secondary Outcome: Percentage of Participants Achieving Objective Response (Objective Response Rate [ORR])
Description: ORR was the percentage of participants with an objective response (complete response [CR] or partial response [PR]). Per RECIST (version 1.1). CR: complete disappearance of all target lesions except nodal disease or disappearance of all non-target lesions and normalization of tumor marker levels. All target nodes/lymph nodes must decrease to normal size (<10 mm short axis); PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions (short diameter=sum for target nodes; longest diameter=sum for all other target lesions). PD: 20% increase in sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm or unequivocal progression of pre-existing non-target lesions or appearance of new unequivocal malignant lesions.
Time Frame: From C1D1 until disease progression or death due to any cause, whichever occurred first (up to maximum of 471 weeks of treatment exposure)
Population: Efficacy analysis set included all enrolled participants who started the treatment of Cycle 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
Percentage of participants | 19.2 [6.6 to 39.4]

29. Secondary Outcome: Percentage of Participants Achieving Disease Control (Disease Control Rate [DCR])
Description: Disease control (DC) = CR, PR or stable disease (SD) >= 24 weeks according to RECIST version 1.1 recorded from C1D1 until disease progression or death due to any cause. CR: complete disappearance of all target lesions except nodal disease or disappearance of all non-target lesions and normalization of tumor marker levels. All target nodes/lymph nodes must decrease to normal size (<10 mm short axis); PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions (short diameter=sum for target nodes; longest diameter=sum for all other target lesions). SD: Does not qualify for CR, PR or progression. PD: 20% increase in sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm or appearance of new unequivocal malignant lesions.
Time Frame: as for outcome 28
Population: Efficacy analysis set included all enrolled participants who started the treatment of Cycle 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
Percentage of participants | 65.4 [44.3 to 82.8]

30. Secondary Outcome: Duration of Response
Description: Duration of response was the time from first documentation of CR or PR to date of first documentation of PD or death for the participants with an objective response (CR or PR). Per RECIST (version 1.1). CR: complete disappearance of all target lesions except nodal disease or disappearance of all non-target lesions and normalization of tumor marker levels. All target nodes/lymph nodes must decrease to normal size (<10 mm short axis); PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions (short diameter=sum for target nodes; longest diameter=sum for all other target lesions). PD: 20% increase in sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm or unequivocal progression of pre-existing non-target lesions or appearance of new unequivocal malignant lesions. Kaplan-Meier method was used.
Time Frame: From first documentation of CR or PR to date of first documentation of objective progression or death, whichever occurred first (up to maximum of 471 weeks of treatment exposure)
Population: Efficacy analysis set included all enrolled participants who started the treatment of Cycle 1. Here, 'Overall Number of Participants Analyzed' signifies participants in the efficacy analysis set who achieved an objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 5
Months | 25.1 [8.3 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of participants with events.

31. Secondary Outcome: 1-Year PFS Probability
Description: PFS was defined as the time from C1D1 to date of first documentation of PD or death due to any cause, whichever occurred first. Documentation of progression was by objective disease assessment as defined by the RECIST (version 1.1). PD was defined as a >=20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 millimeter (mm); or unequivocal progression of pre-existing lesions for non-target disease; or appearance of new unequivocal malignant lesions. One-year PFS probability was defined as the probability (expressed as percentage) of PFS at 1 year after C1D1. PFS probability was determined using the Kaplan-Meier method.
Time Frame: 1 year
Population: Efficacy analysis set included all enrolled participants who started the treatment of Cycle 1.
Measure: Number (95% Confidence Interval); unit: Percentage probability
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
Percentage probability | 57.5 [35.3 to 74.5]

32. Secondary Outcome: Trough Plasma Concentration of Letrozole
Description: Plasma samples were analyzed for letrozole concentrations using a validated, sensitive and specific high-performance liquid chromatography tandem mass spectrometric (HPLC/MS/MS) method.
Time Frame: pre-dose of Cycle 1 Days 19, 20, 21 and Cycle 2 Day 1
Population: "Number of Participants Analyzed" represents all enrolled and treated participants who had letrozole concentration data. "Number Analyzed" represents the number of such participants who had data at each specified time point.
Measure: Median (Full Range); unit: nanograms per milliliter (ng/mL)
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 25
nanograms per milliliter (ng/mL)
  Cycle 1 Day 19 pre-dose: number analyzed (Participants) | 23
  Cycle 1 Day 19 pre-dose | 83.70 [30.8 to 134]
  Cycle 1 Day 20 pre-dose: number analyzed (Participants) | 24
  Cycle 1 Day 20 pre-dose | 83.85 [41.4 to 141]
  Cycle 1 Day 21 pre-dose: number analyzed (Participants) | 24
  Cycle 1 Day 21 pre-dose | 85.30 [38.2 to 134]
  Cycle 2 Day 1 pre-dose | 97.40 [48.8 to 282]

33. Secondary Outcome: Ratio Over Baseline for Skin Biomarker Phosphorylated Retinoblastoma Protein (pRb) Expression
Description: The pRb was one of the skin biomarkers and samples were assayed using immunohistochemistry (IHC) method. Ratio over baseline was calculated by dividing the H-score value for pRb at each specified time point by baseline value. The H-score value, which could range from 0 to 300 (strongest expression) with higher score representing stronger expression, was calculated from the total of each individual intensity of staining (0 [negative], 1+ [weak], 2+ [moderate], 3+ [strong]) multiplied by the percentages of cells (0 to 100) that represented that staining.
Time Frame: Baseline (Day -1), lead-in phase Days 1 and 2, Cycle 1 Days 21, 22, 23, 24, 25, 26
Population: All enrolled and treated participants who had both pre-dose value and at least 1 post dose value for at least 1 biomarker. "Number Analyzed" refers to the number of evaluable participants for each specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
ratio
  Lead-in phase Day 1: number analyzed (Participants) | 12
  Lead-in phase Day 1 | 0.644 (56.34)
  Lead-in phase Day 2: number analyzed (Participants) | 11
  Lead-in phase Day 2 | 0.523 (92.28)
  Cycle 1 Day 21: number analyzed (Participants) | 9
  Cycle 1 Day 21 | 0.535 (108.77)
  Cycle 1 Day 22: number analyzed (Participants) | 11
  Cycle 1 Day 22 | 0.773 (57.77)
  Cycle 1 Day 23: number analyzed (Participants) | 8
  Cycle 1 Day 23 | 0.799 (91.59)
  Cycle 1 Day 24: number analyzed (Participants) | 12
  Cycle 1 Day 24 | 1.493 (103.46)
  Cycle 1 Day 25: number analyzed (Participants) | 9
  Cycle 1 Day 25 | 1.165 (99.39)
  Cycle 1 Day 26: number analyzed (Participants) | 12
  Cycle 1 Day 26 | 2.164 (87.80)

34. Secondary Outcome: Ratio Over Baseline for Skin Biomarker Ki67 Expression
Description: The Ki67 was one of the skin biomarkers and samples were assayed using IHC method. Ratio over baseline was calculated by dividing the percentage of Ki67 positive cells at each specified time point by baseline value.
Time Frame: Baseline (Day -1), lead-in phase Days 1 and 2, Cycle 1 Days 21, 22, 23, 24, 25, 26
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
ratio
  Lead-in phase Day 1: number analyzed (Participants) | 12
  Lead-in phase Day 1 | 0.985 (42.32)
  Lead-in phase Day 2: number analyzed (Participants) | 11
  Lead-in phase Day 2 | 0.868 (64.99)
  Cycle 1 Day 21: number analyzed (Participants) | 9
  Cycle 1 Day 21 | 0.495 (107.24)
  Cycle 1 Day 22: number analyzed (Participants) | 11
  Cycle 1 Day 22 | 0.408 (135.34)
  Cycle 1 Day 23: number analyzed (Participants) | 8
  Cycle 1 Day 23 | 0.599 (80.00)
  Cycle 1 Day 24: number analyzed (Participants) | 12
  Cycle 1 Day 24 | 0.832 (42.34)
  Cycle 1 Day 25: number analyzed (Participants) | 9
  Cycle 1 Day 25 | 0.920 (85.52)
  Cycle 1 Day 26: number analyzed (Participants) | 12
  Cycle 1 Day 26 | 1.301 (61.26)

35. Secondary Outcome: Ratio Over Baseline for Thymidine Kinase (TK) Concentration
Description: Blood samples were collected to provide serum for the assessments of TK activity. The concentrations of TK were determined using enzyme-linked immunosorbent assay (ELISA) method. Ratio of serum TK concentration at each specified time point over baseline value was presented.
Time Frame: Baseline (Day -1 pre-dose), lead-in phase Day 1 (4, 8, 10, 24, 72, 120 hours post dose), Cycle 1 Day 21 (4, 8, 10, 24, 72, 96, 120 hours post dose), Cycle 2 Day 1 pre-dose
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 26
ratio
  Lead-in phase Day 1, 4 hours post dose | 0.780 (44.69)
  Lead-in phase Day 1, 8 hours post dose | 0.774 (43.65)
  Lead-in phase Day 1, 10 hours post dose | 0.733 (49.67)
  Lead-in phase Day 1, 24 hours post dose | 0.702 (48.93)
  Lead-in phase Day 1, 72 hours post dose | 0.530 (50.14)
  Lead-in phase Day 1, 120 hours post dose | 0.598 (74.40)
  Cycle 1 Day 21, 4 hours post dose: number analyzed (Participants) | 23
  Cycle 1 Day 21, 4 hours post dose | 0.260 (172.41)
  Cycle 1 Day 21, 8 hours post dose: number analyzed (Participants) | 23
  Cycle 1 Day 21, 8 hours post dose | 0.236 (191.22)
  Cycle 1 Day 21, 10 hours post dose: number analyzed (Participants) | 23
  Cycle 1 Day 21, 10 hours post dose | 0.236 (187.02)
  Cycle 1 Day 21, 24 hours post dose: number analyzed (Participants) | 24
  Cycle 1 Day 21, 24 hours post dose | 0.247 (164.37)
  Cycle 1 Day 21, 48 hours post dose: number analyzed (Participants) | 24
  Cycle 1 Day 21, 48 hours post dose | 0.244 (166.61)
  Cycle 1 Day 21, 72 hours post dose: number analyzed (Participants) | 24
  Cycle 1 Day 21, 72 hours post dose | 0.268 (163.67)
  Cycle 1 Day 21, 96 hours post dose: number analyzed (Participants) | 24
  Cycle 1 Day 21, 96 hours post dose | 0.292 (176.92)
  Cycle 1 Day 21, 120 hours post dose: number analyzed (Participants) | 24
  Cycle 1 Day 21, 120 hours post dose | 0.455 (334.32)
  Cycle 2 Day 1, pre-dose: number analyzed (Participants) | 24
  Cycle 2 Day 1, pre-dose | 1.069 (248.43)

ADVERSE EVENTS:
Time Frame: From first dose of study medication up to 28 days after last dose of study medication (up to maximum of 475 weeks, maximum treatment exposure = 471 weeks)
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
Groups:
- Palbociclib + Letrozole: Participants received a single dose of palbociclib 125 milligrams (mg) orally on Day 1 during the 5-day lead-in phase and received orally once daily (QD) from Day 1 to Day 21 (followed by 7 days off-treatment) during each 28-day treatment cycle. A treatment cycle was defined as 28 days in duration and Cycle 1 started on Day 6 of lead-in phase as Cycle 1 Day 1. Letrozole 2.5 mg was administered orally QD from Days 1 to 5 during the 5-day lead-in phase and from Days 1 to 28 during each 28-day treatment cycle.
Arm/Group | Palbociclib + Letrozole
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 4/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Letrozole (N=26)
Drug-induced liver injury (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 1
Abscess (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Letrozole (N=26)
Anaemia (Blood and lymphatic system disorders) | 13
Leukopenia (Blood and lymphatic system disorders) | 11
Neutropenia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Sinus tachycardia (Cardiac disorders) | 2
Lenticular opacities (Eye disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Gingival pain (Gastrointestinal disorders) | 2
Gingival ulceration (Gastrointestinal disorders) | 4
Mouth ulceration (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 5
Pyrexia (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 11
Blood alkaline phosphatase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 3
Blood creatinine increased (Investigations) | 2
Blood glucose increased (Investigations) | 3
Blood insulin increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 4
Haemoglobin decreased (Investigations) | 6
Low density lipoprotein increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 16
Platelet count decreased (Investigations) | 15
Red blood cell count decreased (Investigations) | 3
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 4
White blood cell count decreased (Investigations) | 15
Decreased appetite (Metabolism and nutrition disorders) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT02499146/Prot_002.pdf
  • Statistical Analysis Plan (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT02499146/SAP_003.pdf